CLINICAL TRIAL: NCT00972673
Title: Phase I Study of GW685698X-A Randomized, Double Blind, Placebo Controlled, Parallel-group, Repeat Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled Dose From a Novel Dry Powder Device in Healthy Japanese Male Subjects.
Brief Title: A Study of GW685698X in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 112018
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- arm 1 (Experimental): In Arm 1 subjects will receive 200, 400 or 800 microgram of powdered inhalation of GW685698X once daily for 7 days from Day 5 to Day 11.
  Interventions: Drug: GW685698X
- arm 2 (Placebo Comparator): In Arm 2 subjects will receive Placebo powdered inhalation once daily for 7 days from Day 5 to Day 11.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — comparator
  Arms: arm 2
Drug: GW685698X — Inhaled steroid
  Arms: arm 1

SUMMARY:
This is a randomized, double blind, placebo controlled, parallel-group, repeat dose study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of inhaled dose from a novel dry powder device in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy male subjects aged between 20 and 64 years of age inclusive. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination, laboratory studies, and other tests.
* Body weight ≥ 50kg and BMI within the range 18.5-25.0kg/m2 inclusive.
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked))
* Clinical laboratory tests data obtained at screening meet the following:

AST(GOT), ALT(GPT), total-bilirubin: below the upper limit of the normal ranges

* Normal 12-lead EGC finding at screening; QTc(B) interval <450msec
* Normal spirometry (FEV1 ≥ 80% of predicted, FEV1/FVC ≥ 70%).
* Rapid ACTH with normal range at the screening.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Capable of using the novel dry powder inhaler.

Exclusion Criteria:

* The subject has any clinically relevant abnormality on medical examination, vital sign, clinical laboratory test or medical history at screening in the medical opinion of the investigator or the subject has a medical history that is not considered as eligible for inclusion in this study by the investigator.
* The subject has an allergy for any drug or idiosyncrasy
* The subject has an allergy for any drug hypersensitivity to milk protein or the excipients lactose monohydrate and magnesium stearate.
* T he subject is currently participating in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
* The subject has participated in a clinical study with an investigational or a non-investigational drug or device during the previous 4 months.
* The subject has a history or current conditions of drug abuse or alcoholism.
* History of regular alcohol consumption exceeding on average, 14 drinks/week (1 drink = 5 ounces (150mL) of wine or 350mL of beer or 1.5 ounces (45mL) of 80 proof distilled spirits) within 6 month of screening.
* The subject is positive for urine drug at screening.
* Use of prescription or non-prescription drugs, including CYP3A/PGP inhibitor, vitamins, herbal and dietary supplements (including St John'sWort) within 14 days prior to the first dose of study medication.
* The subject has a known allergy or hypersensitivity to corticosteroids.
* The subject has a known allergy or hypersensitivity to synthetic ACTH
* The subject has a history of asthma in childhood or respiratory disorder.
* The subject is a permanent (or occasional during the study) night-shift worker*.

  * Permanent night shift worker defines as the person who has been continuing life that gets up after 12:00 day time and eats supper after 0:00 midnight for seven days or more usually.
* The subject is positive for syphilis, HBs antigen, HCV antibody, HIV antibody, HTLV-1 antibody.
* The subject has donated a unit of blood ">400mL" within the previous 4 months or ">200mL" within the previous 1 month.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-09-24 (Actual); Primary Completion 2008-12-19 (Actual); Study Completion 2008-12-19 (Actual)

PRIMARY OUTCOMES:
safety: adverse events, vital sign, ECGs, and clinical laboratory test
PK： Cmax, tmax and AUC(0-t)
PD: serum cortisol

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Kagoshima, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Nakahara N, Wakamatsu A, Kempsford R, Allen A, Yamada M, Nohda S, Hirama T. The safety, pharmacokinetics and pharmacodynamics of a combination of fluticasone furoate and vilanterol in healthy Japanese subjects. Int J Clin Pharmacol Ther. 2013 Aug;51(8):660-71. doi: 10.5414/CP201822. PMID 23735179
- See also: Results for study 112018 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112018?search=study&search_terms=112018#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112018 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112018 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112018 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112018 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register